CLINICAL TRIAL: NCT04227795
Title: Artificial Intelligence-Assisted Real-time Detection of Missed Lesions During Colonoscopy: A Prospective Study
Brief Title: AI-assisted Detection of Missed Colonic Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, LEUNG Wai Keung, Clinical Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UW 19-309
Record Dates: First submitted 2020-01-10; First posted 2020-01-14 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Colon Adenoma; Colonic Polyp; Colon Cancer
Keywords: Artificial intelligence; Colonoscopy; Deep learning; Detection; Computer-aided
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificial intelligence-Assisted real time colonoscopy (Experimental): AI assisted real-time detection of colonic lesions
  Interventions: Device: Artificial intelligence-Assisted real time colonoscopy

INTERVENTIONS:
Device: Artificial intelligence-Assisted real time colonoscopy — The colonoscopy was performed under artificial intelligence assistance

SUMMARY:
A prospective validation of real time deep learning artificial intelligence model for detection of missed colonic polyps

DETAILED DESCRIPTION:
Consecutive adult patients, age 40 or above, who were scheduled to have outpatient colonoscopy in the Queen Mary Hospital were invited to participate. Patients were excluded if they were unable to provide informed consent, considered to be unsafe for taking biopsy or polypectomy including patients with bleeding tendency and those with severe comorbid illnesses. Also, patients with history of inflammatory bowel disease, familial adenomatous polyposis, Peutz-Jeghers syndrome or other polyposis syndromes were excluded.

The primary endoscopist conducted the colonoscopic examination in the usual manner. All colonoscopy procedures were performed with high-definition colonoscopes (EVIS-EXERA 290 video system, Olympus Optical, Tokyo, Japan). The colonoscopy was first advanced to the cecum in all patients as confirmed by identification of the appendiceal orifice and ileocecal valve or by intubation of the ileum. After cecal intubation, the colonoscopy was slowly withdrawn to the rectum by the primary endoscopist. The AI real time detection was then activated with the output displayed in a different monitor and was only viewed by an independent investigator, who was an experienced endoscopist. The primary endoscopist was blinded to the AI real time detection result al.

The colon was divided into three segments during the examination: right side, transverse and left side colon, using hepatic flexure and splenic flexure as dividing landmark. All polyps were marked for size (measured with biopsy forceps), location and morphology according to the Paris classification, and then removed or biopsied for histological examination. After examination of each segment, segmental unblinding of the AI results were provided by the independent viewer. If additional polyps were detected by AI but not by the endoscopist, that segment were reexamined to look for the missed polyp. If no additional polyp was detected by the AI, the next colonic segment was examined. Missed lesions were defined as lesions identified by AI and then confirmed on reexamination by the endoscopist.

The first withdrawal time (minus the polypectomy site) was measured. The Boston Bowel Preparation Scale score (BPPS) was used for evaluation of bowel cleanliness.

ELIGIBILITY:
Inclusion Criteria:

* consecutive adult patients, age 40 or above, who were scheduled to have outpatient colonoscopy in the Queen Mary Hospital were invited to participate

Exclusion Criteria:

* Patients were excluded if they were unable to provide informed consent, considered to be unsafe for taking biopsy or polypectomy including patients with bleeding tendency and those with severe comorbid illnesses.
* Also, patients with history of inflammatory bowel disease, familial adenomatous polyposis, Peutz-Jeghers syndrome or other polyposis syndromes were excluded.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Adenoma miss rate | During the colonoscopy procedure
  The number of patient had at least one missed adenoma

SECONDARY OUTCOMES:
Total number of adenoma missed | During the colonoscopy procedure
  The total number of missed polyps for all subjects
Colonic polyp miss rate | During the colonoscopy procedure
  The number of patient had at least one missed adenoma
Total number of missed polyps | During the colonoscopy procedure
  The total number of missed polyps for all subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ka Luen, Thomas Lui, Principal Investigator — Queen Mary Hospital, the University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lui TKL, Hui CKY, Tsui VWM, Cheung KS, Ko MKL, Foo DCC, Mak LY, Yeung CK, Lui TH, Wong SY, Leung WK. New insights on missed colonic lesions during colonoscopy through artificial intelligence-assisted real-time detection (with video). Gastrointest Endosc. 2021 Jan;93(1):193-200.e1. doi: 10.1016/j.gie.2020.04.066. Epub 2020 May 4. PMID 32376335